CLINICAL TRIAL: NCT01838759
Title: Bioimpedance Spectroscopy for the Differential Diagnosis of Hyponatremia
Status: Completed | Type: Observational
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Ender Hur, Associate Professor Doctor, Zonguldak Bulent Ecevit University
Other Study IDs: BEUN 2013-31-26/02
Record Dates: First submitted 2013-04-20; First posted 2013-04-24 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Hyponatremia
Keywords: Bioimpedance spectroscopy; Hypervolemia; Hypovolemia
MeSH Terms: conditions — Hyponatremia; Edema; Hypovolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hypovolemic hyponatremia: Negative values of "Overhydration" measured by Bioimpedance spectroscopy
- Hypervolemic hyponatremia: Positive values of "Overhydration" measured by Bioimpedance spectroscopy

SUMMARY:
We aimed to investigate the role of bioimpedance spectroscopy for the diagnosis of hyponatremia

DETAILED DESCRIPTION:
* Up to now, "Hyponatremia" differentially diagnosed by physical examination, plasma and urine osmolalities, Echocardiography and biochemical measurements.
* The purpose of this study is to determine whether bioimpedance spectroscopy can be used for the detection of hypovolemia and hypervolemia for the differential diagnosis of hyponatremia.

ELIGIBILITY:
Inclusion Criteria:

* Willing to participate in the study with written informed consent
* Older than 18-years

Exclusion Criteria:

* The presence of pacemaker or defibrillator
* Artificial joints, pin or amputation
* Pregnancy or lactating.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Bulent Ecevit University Hospital with the presentation of hyponatremia
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2013-02; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Accuracy of volume status measured by bioimpedance spectroscopy | Six months
  BIOIMPEDANCE SPECTROSCOPY:
  Overhydration (OH) measurement by Body Composition Monitor (Fresenius Medical Care)
  Negative values of "OH" indicating Hypovolemia and positive values for hypervolemia in hyponatremic patients.

SECONDARY OUTCOMES:
Laboratory data and echocardiography | 6 Months
  LABORATORY MEASUREMENTS Hemoglobin, Hematocrit, White blood cell count Platelet count, Na, Potassium, Chlorur, Urea, Creatinine, Uric acid, Plasma osmolality, Urine osmolality, Alanine transaminase , Aspartate transaminase , Urine specific gravity,
  TREATMENT MODALITY
  1. Diuretics
  2. Intravenous hydration by isotonic saline
  ECHOCARDIOGRAPHY:
  Left ventricular end-diastolic diameter, Left ventricular end-systolic diameter, Ejection fraction(%), Left Atrium diameter, Aortic diameter, Right atrium diameter, Interventricular septum, Posterior wall thickness, Mitral insufficiency, Pulmonary insufficiency, Systolic pulmonary artery pressure, Tricuspid insufficiency

CONTACTS AND LOCATIONS:
Overall Officials: Ender Hur, Assoc.Prof., Study Chair — Bulent Ecevit University Medical School, Division of Nephrology, Zonguldak, Turkey
Locations (1):
- Bulent Ecevit University Hospital, Zonguldak, Turkey (Türkiye)

REFERENCES:
- [Background] Hur E, Usta M, Toz H, Asci G, Wabel P, Kahvecioglu S, Kayikcioglu M, Demirci MS, Ozkahya M, Duman S, Ok E. Effect of fluid management guided by bioimpedance spectroscopy on cardiovascular parameters in hemodialysis patients: a randomized controlled trial. Am J Kidney Dis. 2013 Jun;61(6):957-65. doi: 10.1053/j.ajkd.2012.12.017. Epub 2013 Feb 15. PMID 23415416
- [Derived] Kose SB, Hur E, Magden K, Yildiz G, Colak D, Kucuk E, Toka B, Kucuk H, Yildirim I, Kokturk F, Duman S. Bioimpedance spectroscopy for the differential diagnosis of hyponatremia. Ren Fail. 2015 Jul;37(6):947-50. doi: 10.3109/0886022X.2015.1040418. Epub 2015 Apr 27. PMID 25915455